CLINICAL TRIAL: NCT00589368
Title: Interhemispheric Transfer of Grasp Control After Stroke
Brief Title: Transfer of Grasp Control Across Hands After Stroke
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Preeti Raghavan, Assistant Professor of Rehabilitation Medicine, NYU Langone Health
Other Study IDs: 04-0585; K23HD049472 (NIH)
Record Dates: First submitted 2007-12-24; First posted 2008-01-09 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Stroke With Hemiparesis
Keywords: Brain Infarction; pathology; physiopathology; psychology; rehabilitation; Fingers; Grasp; Functional Laterality; Hand; Strength; Neuronal Plasticity; Psychomotor Performance; Biomechanis; Touch; Weight-Bearing
MeSH Terms: conditions — Brain Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: stroke group
  Interventions: Behavioral: Transfer of grasp control across hands
- 2: control group
  Interventions: Behavioral: Transfer of grasp control across hands

INTERVENTIONS:
Behavioral: Transfer of grasp control across hands — transfer of planning and execution of grasp across hands in terms of its effect on fingertip forces, and the timing and magnitude of muscle contraction in patients with hemiparesis and healthy controls

SUMMARY:
The purpose of this study is to examine if the strong hand can assist in the recovery of muscle function in the weak hand after a stroke.

DETAILED DESCRIPTION:
Hemiparesis is the most common motor impairment after stroke. Persistent deficits in the distal upper extremity lead to impaired hand function and disability in Activities of Daily Living, accruing enormous costs in terms of health care services and lost productivity. The mechanisms of recovery of hand motor function after stroke are poorly understood, and the protocols used in clinical practice lack a solid scientific rationale. Prior work has shown that grasping with the non-involved hand may assist in planning of grasp with the involved hand after stroke. The goal of the proposed project is to investigate the type and nature of information relayed across the hemispheres by prior manipulation with the non-involved hand to improve planning and control of grasp with the involved hand. Psychophysical methods using a grip instrument will be used to examine the type of information necessary for planning of grasp, and quantitative surface electromyography will be used to investigate the contribution of improved planning to neuromuscular control of grasp. Integration of these methods in the study of grasp control will clarify the neural mechanisms underlying hand dysfunction, and facilitate the development of rational therapeutic protocols for upper extremity rehabilitation after stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Previously right-handed subjects with hemiparesis and complaints of unilateral hand dysfunction during grasping resulting from a single unilateral cerebral infarct in the MCA territory affecting either the right or the left side of the brain at least 3 months prior to data collection
2. Previously right-handed healthy control subjects age-matched to the stroke patients
3. All subjects must have the ability to reach, grasp and lift the test object with both extremities (stroke patients with the impaired extremity as well) and complete the experimental protocol as assessed by the PI.
4. All subjects must score > 24 on the Folstein's mini-mental exam to screen out significant cognitive dysfunction
5. Subjects must obtain MRI or CT scan images of their brain taken since their stroke, or be willing to have a structural MRI or CT scan taken as part of this research study.

Exclusion Criteria:

1. Presence of clinically significant visual deficits, aphasia, neglect, or apraxia as determined by clinical neurologic examination that may interfere with the research protocol
2. Presence of sensory deficits in control subjects and in the non-involved hand of stroke subjects on testing of two-point discrimination
3. History of surgery or other significant injury to the upper extremities
4. Botulinum toxin injections in the upper extremity musculature in the three months prior to enrollment in the study.
5. Current treatment with intrathecal baclofen
6. Previous neurological illness such as head trauma, prior stroke, epilepsy, demyelinating disease
7. Complicating medical problems such as uncontrolled, diabetes with polyneuropathy, severe renal, cardiac or pulmonary disease, or any other severe concurrent medical problem that will interfere with obtaining reliable results.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with stroke will be recruited from the inpatient and outpatient Rehabilitation units at the Mount Sinai Medical Center and from referrals by community rehabilitation physicians and neurologists. Control subjects will be recruited by public advertisement in the New York City area. There are no exclusions based on gender or ethnic groups.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2006-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Difference in peak load force rates for grasping a light and a heavy weight object as measured using a custom made object with 6 dof force sensors. | immediately post-intervention

SECONDARY OUTCOMES:
Timing and magnitude of motor unit recruitment as measured by quantitative EMG of the grasping and lifting muscles. | immediately post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Raghavan, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- Rusk Institute of Rehabilitation Medicine, New York, New York, United States